CLINICAL TRIAL: NCT06893471
Title: From Annual Measurements to Daily Improvements: Evaluation of a Method for Improving Systematic Work Environment Management
Brief Title: From Yearly Checks to Daily Progress: Evaluating Goal Attainment Scaling (GAS) in Systematic Work Environment Management (SAM) Within the Municipal Sector
Acronym: GAS for SAM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Mälardalen University (Other)
Responsible Party: Principal Investigator, Sebastian Heikklä, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20240063 (AFA-grant); 20240063 (Other Grant/Funding Number: AFA-insurance)
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Behavior Change Interventions; Work Environment Adverse Effects; Health Factors; Goal Attainment Scaling
Keywords: Goal Attainment Scaling (GAS); Systematic work engagement management (SAM); group level; municipal sector; goal setting; RCT; health factors; Step Wedge Design
MeSH Terms: conditions — Occupational Stress | interventions — S-Adenosylmethionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Business-as-usual condition: This group follows established processes for systematic work engagement management (SAM)
  We will employ a randomization approach using a two-arm stepped-wedge design. This design allows for a sequential roll-out of the intervention across study arms while maintaining a randomized allocation schedule. The stepped-wedge approach ensures that all participants eventually receive the intervention, while still permitting valid between-group comparisons at different time points. Importantly, this design also enables the inclusion of an additional measurement point, which will strengthen our ability to assess both short-term and longer-term intervention effects.
- Experiment group (Experimental): Works with Goal Attainment Scaling (GAS) as part of systematic work engagement management (SAM)
  We will employ a randomization approach using a two-arm stepped-wedge design. This design allows for a sequential roll-out of the intervention across study arms while maintaining a randomized allocation schedule. The stepped-wedge approach ensures that all participants eventually receive the intervention, while still permitting valid between-group comparisons at different time points. Importantly, this design also enables the inclusion of an additional measurement point, which will strengthen our ability to assess both short-term and longer-term intervention effects.
  Interventions: Other: GAS for SAM

INTERVENTIONS:
Other: GAS for SAM — This study adapts Goal Attainment Scaling (GAS) for group-level goal setting within systematic work environment management. Developed collaboratively with organizational stakeholders, the method is:
  Tailormade - Allows flexibility in defining and scaling goals. Co-created - Encourages ownership and employee involvement. Standardized - Uses a five-level scale (-2 to +2) for tracking progress and enabling comparisons.
  Data-driven - Includes a Progress Graph for systematic follow-up and documentation of goals and initiatives.
  Managers in the experiment group will receive training before implementation begins
  Arms: Experiment group

SUMMARY:
The goal of this project is to evaluate a practical method for improving systematic work environment management (SAM) by focusing on health-promoting factors rather than identifying risk-factors, and deficiencies. It will also explore how Goal Attainment Scaling (GAS) can support goal-setting and evaluation within SAM. The main questions it aims to answer are:

* Which health-promoting factors are prioritized, and what organizational-level initiatives are developed?
* How does using GAS influence goal achievement related to health-promoting factors?
* How do employees, managers, and HR representatives perceive the use of GAS?
* What factors help or hinder the implementation of GAS and goal attainment?

Participants will:

Apply GAS within their organizations to set and evaluate goals Engage in a participatory process to identify key health-promoting factors Assess progress and the impact of interventions over time Researchers will analyze the effectiveness of GAS in enhancing SAM (experiment vs control group) and develop tools to support sustainable, healthy workplaces in the municipal sector.

DETAILED DESCRIPTION:
This project aims to test and evaluate a practical method for enhancing systematic work environment management (SAM), shifting the focus from identifying deficiencies to achieving goals centered on health-promoting factors. Competence supply is one of the greatest challenges for Swedish municipalities, and deficiencies in organizational and social work environments contribute significantly to sickness absence, poor mental health, and well-being. This issue threatens municipalities' ability to fulfill their responsibilities to citizens. Active systematic work environment management (SAM) has been identified as a potential solution, yet many municipalities rely on annual assessments focused on shortcomings, without providing indicators for concrete solutions, goal achievement, or measurable progress.

There is a lack of knowledge on how SAM should be designed to prioritize health-promoting factors (i.e., workplace conditions that support employee health and sustainable employment) at an organizational level. Additionally, there is a need for goal indicators that are motivating, measurable, and applicable at both unit and organizational levels.

To address these pressing needs, we propose applying the Goal Attainment Scaling (GAS) method. GAS serves as both a goal-setting and evaluation methodology, previously applied successfully at the individual level. We suggest that GAS can help organizations formulate concrete and tailored desired states related to specific interventions, thereby enhancing improvements in health-promoting factors.

GAS offers several advantages for enhancing SAM. First, goal-setting theory suggests that GAS facilitates the establishment of achievable and relevant goals. A participatory design is crucial, fostering a shared mental model of objectives. Second, GAS promotes data-driven decision-making and accountability within SAM, enabling workplaces to systematically assess progress and the impact of work environment initiatives. Third, GAS is versatile and universal, serving as a general framework adaptable to different organizations and their specific contexts and objectives.

The project will address the following research questions:

1. Which health-promoting factors are prioritized, and what organizational-level initiatives are generated to address them?
2. How does the application of GAS (as part of SAM) influence the achievement of goals related to health-promoting factors?
3. How is the use of GAS perceived by different stakeholders (employees, managers, HR representatives)?
4. What facilitators and barriers influence the implementation of GAS and the attainment of goals? The project will identify and highlight prioritized organizational-level health-promoting factors while mapping successful strategies and practices for addressing them. The expected outcome is the development of a systematic, participatory, and practical method that fosters local engagement in initiative development, goal setting, and follow-up of health-promoting factors within SAM. This work will contribute to the development of measurement methods and outcome metrics for organizational-level health-promoting factors. The resulting knowledge and tools can support the creation of long-term healthy, sustainable, and attractive workplaces within the municipal sector

ELIGIBILITY:
Inclusion Criteria:

* work unit must have >3 employees, working within municipal sector, no other major organizational changes

Exclusion Criteria:

* Units with <3 employees, other major organizational changes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Employee survey results | From enrollment to the end of treatment at 2 years
  The results from the annual employee survey will be the primary outcome in this study.
  The municipality uses e.g., HME index from Sveriges Kommuner och Regioner (SKR) and are developing specific items for measuring health factors built on research based questions.
  1. Fair and transparent organization:
     Colquitt, 2001; COPSOQIII; Rawlins, 2008
  2. Leadership (present, trusting, engaging):
     Carless et al. 2000
  3. Participation and influence:
     Astvik et al. 2020; QPS Nordic
  4. Communication and feedback:
     Astvik et al. 2020
  5. Prioritization of work tasks:
     Astvik et al. 2020; COPSOQIII; Semmer et al. 2007; Åkerblom et al. 2021
  6. Lifelong competence development:
     COPSOQIII; Singer et al. 2012; OSA
  7. Systematic work environment management in daily practice:
     Berthelsen et al. 2020
  8. Early interventions and work adjustments:
  COPSOQIII
  Responses are rated on a five point (1-5) Likert-scale (higher score better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrica von Thiele Schwarz, Professor in Psychology, Study Chair — Mälardalen University
Locations (1):
- Hudiksvall municipality, Hudiksvall, Gävleborg County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This is a collaborative project with a municipality. Data will be collected at the group level (work units) and will remain confidential.